CLINICAL TRIAL: NCT05862467
Title: Efficacy of a Posttraumatic Stress Disorder (PTSD) Intervention for Autistic Adults on Biobehavioral Health
Brief Title: A Pilot Participatory Program Evaluation of a Virtual Trauma Support Program for Autistic Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wyoming (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20230331CM03524
Record Dates: First submitted 2023-04-25; First posted 2023-05-17 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Autism; Trauma; Posttraumatic Stress Disorder; Posttraumatic Stress Symptom
MeSH Terms: conditions — Autistic Disorder; Wounds and Injuries; Stress Disorders, Post-Traumatic | interventions — Wettability

STUDY DESIGN:
Intervention Model Description: This is a single group study, where all participants receive telehealth-based Written Exposure therapy (WET). Feasibility and initial efficacy is assessed via pre-post assessments, conducted pre-WET, at the end of WET, and 1 and 6 months post program completion.
Masking Description: No masking -- as single group design, all participants receive the program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Written Exposure Therapy (Experimental): Behavioral therapy: Written Exposure Therapy via telehealth
  Interventions: Behavioral: Written Exposure Therapy (WET) via telehealth

INTERVENTIONS:
Behavioral: Written Exposure Therapy (WET) via telehealth — Written Exposure Therapy (WET) via telehealth

SUMMARY:
The goal of this single-group clinical trial is to learn about the initial efficacy and feasibility of telehealth-delivered Written Exposure Therapy (WET) for autistic adults with traumatic stress symptoms. The main questions the investigators aim to answer are:

* Do symptoms of posttraumatic stress disorder (PTSD) and co-occurring mental health concerns decrease after receiving WET?
* Do biobehavioral health outcomes, including objective (Fitbit indicators of activity, sleep, and heart rate) and subjectively-reported health variables (e.g., sleep, pain, health-related quality of life), improve after receiving WET?
* How do autistic adults experience WET, and how can this program be modified and enhance in the future in collaboration with autistic adults?

Participants will complete the following as part of the study, which is completed entirely over telehealth.

* Participants will first complete an initial assessment, involving brief measures of cognition and autistic traits, as well as interviews and questionnaires about PTSD, mental health, and physical health. If eligible, participants will proceed to the following steps:
* Eligible participants will then start wearing a Fitbit, to be used for the duration of the study.
* Participants will then participate in 5 weekly virtual visits involving the WET protocol, including weekly brief assessment of PTSD and mental and physical health.
* Then, participants will complete a sixth virtual visit the following week where PTSD, mental and physical health, and treatment feedback are assessed.
* Lastly, participants will complete virtual visits 1 and 6 months later involving re-assessment of PTSD and mental and physical health.

Therefore, this is a pre-post single group design, where all participants will receive WET to establish initial efficacy and feasibility. Investigators will also consult with an autistic advisory board throughout the project, and make adaptations as recommended in consultation with autistic adults. The goal is to better understand the initial efficacy and feasibility of WET for supporting autistic adults who have experienced trauma.

ELIGIBILITY:
Inclusion Criteria:

* Autistic
* Age 18 years or over
* Has experienced trauma and reports clinically significant symptoms of traumatic stress (clinically elevated score on either Posttraumatic Symptom Checklist (PCL-5) or Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders (SCID-5), and/or other self-report/interview evidence of significant traumatic stress symptoms for which participant wants support/program
* Comfortable speaking and writing in English
* Full Scale Intelligence Quotient (FSIQ) score >= 65 (given written nature of Written Exposure Therapy) on the Wechsler Abbreviated Scale of Intelligence-Second Edition (WASI-2)
* Access to device with internet access for telehealth visits

Exclusion Criteria:

* Participant is not Autistic
* Participant is unable to understand English
* Participant is currently receiving trauma-focused therapeutic services
* Participant does not have access to internet connected device for telehealth visits
* Participant receives Full Scale Intelligence Quotient (FSIQ) score < 65 on the Wechsler Abbreviated Scale of Intelligence-Second Edition (WASI-2)
* If there are significant safety concerns for any participant (e.g., imminent risk of harm to self or other) the Principal Investigator may determine whether it is not in the adult's best interest to be enrolled given that this study does not provide care/services relating to active risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-10-26 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
Change in posttraumatic stress disorder (PTSD) symptoms on the Posttraumatic Symptom Checklist for DSM-5 (PCL-5) Scale | Change across baseline to follow-up (an average of 6 months)
  The Posttraumatic Symptom Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 is a self-report questionnaire of posttraumatic stress disorder symptoms. Total scores range from 0-80; higher scores indicate higher levels of posttraumatic stress disorder symptoms.

SECONDARY OUTCOMES:
Change in depressive symptoms on the Patient Health Questionnaire (PHQ) Scale | Change across baseline to follow-up (an average of 6 months)
  The PHQ is a self-report measure of depressive symptoms. Total scores range from 0-27; higher scores reflect greater levels of depressive symptoms.
Change in anxiety symptoms on the Anxiety Scale for Autism-Adults (ASA-A) | Change across baseline to follow-up (an average of 6 months)
  The Anxiety Scale for Autism-Adults (ASA-A) is a self-report measure for anxiety symptoms among autistic adults. Total scores range from 0 to 60; higher scores reflect higher anxiety symptoms. Three subscales are also scored: social anxiety, anxious arousal, and uncertainty.
Change in loneliness symptoms on the University of California Los Angeles (UCLA) 3-Item Loneliness Scale | Change across baseline to follow-up (an average of 6 months)
  The University of California Los Angeles (UCLA) 3-Item Loneliness Scale is a self-report measure for symptoms of loneliness. Scores range from 3 to 9; higher scores reflect higher levels of loneliness.
Change in psychological adjustment concerns on the Brief Adjustment Scale (BASE-6) | Change across baseline to follow-up (an average of 6 months)
  The Brief Adjustment Scale (BASE-6) is a brief self-report symptom monitoring measure for general psychological adjustment. Scores from from 6 to 42; higher scores reflect greater psychological adjustment concerns.
Change in experiential avoidance symptoms on the Brief Experiential Avoidance Questionnaire | Change across baseline to follow-up (an average of 6 months)
  The Brief Experiential Avoidance Questionnaire is a self-report measure of experiential avoidance. Scores range from 15 to 90; higher scores reflect greater levels of experiential avoidance.
Change in emotion regulation difficulties on the Difficulties in Emotion Regulation Scale (DERS-16) | Change across baseline to follow-up (an average of 6 months)
  The Difficulties in Emotion Regulation Scale (DERS-16) is a self-report measure of emotion regulation difficulties. Scores range from 16 to 80; higher scores reflect greater emotion regulation difficulties.
Change in stigma towards help-seeking on the Ultra-Brief Self-Stigma of Seeking Help (SSOSH-3) Scale | Change across baseline to follow-up (an average of 6 months)
  The Ultra Brief Self-Stigma of Seeking Help (SSOSH-3) Scale is a self-report measure of stigma towards seeking psychological support. Scores range from 3 to 15; higher scores reflect greater stigma.
Change in camouflaging on the Camouflaging Autistic Traits Questionnaire (CATQ) | Change across baseline to follow-up (an average of 6 months)
  The Camouflaging Autistic Traits Questionnaire (CATQ) is a self-report measure of masking autistic traits. Scores range from 25 to 175; greater scores reflect a higher level of camouflaging. Three subscales are scored: Assimilation, Compensation, and Masking.
Change in sleep difficulties on the Pittsburgh Sleep Quality Index (PSQI) | Change across baseline to follow-up (an average of 6 months)
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report measure of sleep difficulties. Scores range from 0 to 21; higher scores reflect greater sleep difficulties.
Change in pain intensity on the Patient-Reported Outcome Measurement Information System (PROMIS) Pain Intensity Short Form Scale. | Change across baseline to follow-up (an average of 6 months)
  The Patient-Reported Outcome Measurement Information System (PROMIS) Pain Intensity Short Form Scale is a self-report measure of pain intensity. Total scores range from 3 to 15; higher scores reflect more intense pain.
Change in pain interference on the Patient-Reported Outcome Measurement Information System (PROMIS) Pain Interference Short Form Scale. | Change across baseline to follow-up (an average of 6 months)
  The Patient-Reported Outcome Measurement Information System (PROMIS) Pain Interference Short Form Scale is a self-report measure of pain interference. Total scores range from 8 to 40; higher scores reflect a greater level of pain interference.
Change in health-related quality of life on the Centers for Disease Control Health-Related Quality of Life Scale (CDC HRQOL) | Change across baseline to follow-up (an average of 6 months)
  The Centers for Disease Control Health-Related Quality of Life Scale (CDC HRQOL) is a self-report of health-related quality of life (CDC HRQOL). The measure yields a number of unhealthy days (from 0 to 30); higher numbers reflect worse health-related quality of life.
Change in PTSD symptoms on the clinician-administered Structured Clinical Interview for DSM-5 | Change across baseline to follow-up (an average of 6 months)
  The Structured Clinical Interview for Diagnostic and Statistical Manual for Mental Disorders (DSM)-5 (SCID-5) is a clinical interview for symptoms of mental health diagnoses. The measure yields number of symptoms for which an individual meets criteria, and whether an individual meets diagnostic criteria, indicating that the person experiences a clinically significant amount of mental health symptom in a particular domain. The PTSD symptom module will be used.
Change in physical activity as assessed on Fitbit. | Change across baseline to follow-up (an average of 6 months)
  Participants Fitbit measurements of number of steps will be assessed via their Fitbit device. A higher number of steps indicates a higher level of physical activity.
Change in sleep quality as assessed on Fitbit. | Change across baseline to follow-up (an average of 6 months)
  Participants Fitbit measurements of sleep quality will be assessed via their Fitbit device. A higher sleep quality indicates overall better sleep outcomes.
Change in sleep duration as assessed on Fitbit. | Change across baseline to follow-up (an average of 6 months)
  Participants Fitbit measurements of sleep duration in hours will be assessed via their Fitbit device. A higher sleep duration indicates greater numbers slept.
Change in resting heart rate as assessed on Fitbit. | Change across baseline to follow-up (an average of 6 months)
  Participants Fitbit measurements of resting heart rate will be assessed via their Fitbit device. Lower resting heart rate indicates a more positive health outcome.

OTHER OUTCOMES:
Change in autistic quality of life on the Autism Spectrum Quality of Life Scale. | Change across baseline to follow-up (an average of 6 months)
  The Autism Spectrum Quality of Life Scale is a self-report measure of quality of life relating to autism. Higher scores reflect greater quality of life.
Change in overall quality of life on the World Health Organization Quality of Life Scale | Change across baseline to follow-up (an average of 6 months)
  The World Health Organization Quality of Life Scale (WHO QOL) is a 26-item self-report questionnaire of quality of life. Higher scores reflect greater quality of life.
Change in positive Autistic identity on the Autism Spectrum Identity Scale (ASIS) | Change across baseline to follow-up (an average of 6 months)
  The Autism Spectrum Identity Scale (ASIS) is a 22-item self-report of autistic identity; higher scores reflect a more positive Autistic identity.
End of program working alliance reported on the Working Alliance Inventory (Short-Revised) | 6 weeks (after baseline, on average)
  The Working Alliance Inventory is a self-report measure of therapeutic alliance. Scores range from 12 to 60; higher scores reflect a greater therapeutic alliance.
End of program satisfaction reported on the Program Satisfaction Questionnaire | 6 weeks (after baseline, on average)
  The Program Satisfaction Questionnaire assesses satisfaction with various aspects of the program.
History of benevolent/positive childhood experiences reported on the Benevolent Childhood Experiences Checklist. | Baseline
  The Benevolent Childhood Experiences checklist is a measure of 20 benevolent/positive childhood experiences. Scores range from 0-20; higher scores reflect greater positive childhood experiences.
History of adverse experiences on the Sexual and Gender Minority Adverse Childhood Experiences Scale | Baseline
  The Sexual and Gender Minority Adverse Childhood Experiences Scale (SGM-ACEs) contains 7 items rated as present or not, and on a scale from never to always. Total scores range from 0 to 35; higher scores reflect a greater frequency of adverse experiences.
Racial trauma symptoms on the Racial Trauma Scale (RTS-Brief Research Version) | Baseline
  The Racial Trauma Scale is a self-report measure of racial trauma symptoms. Scores range from 9 to 36; higher scores reflect a higher level of symptoms. Subscales for lack of safety, negative cognitions, and difficulty coping are scored.
Discrimination experiences on the Everyday Discrimination Scale (EDS) | Baseline
  The Everyday Discrimination Scale (EDS) is a 9-item scale of experiences of discrimination. Scores range from 0 to 45; greater scores indicate more experiences of discrimination.
History of childhood stressful experiences on the Childhood Experiences Survey | Baseline
  The Childhood Experiences Survey is a 17-item measure that assesses the frequency of stressful childhood experiences. Higher scores reflect a greater frequency of stressful experiences.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wyoming, Laramie, Wyoming, United States

IPD SHARING:
Plan to Share IPD: No